CLINICAL TRIAL: NCT00584688
Title: A Double Blind, Placebo Controlled Trial of Quetiapine in Anorexia Nervosa, a Dual Site Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: University of South Florida (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 0825
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2009-03

CONDITIONS: Anorexia Nervosa
Keywords: anorexia; nervosa; eating; disorder; study; research; clinical; trial; psychiatry; psychiatric
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Disease | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: quetiapine — quetiapine dosage will be titrated to subject tolerance beginning at 50 mg every 24 hours upwards to 400 mg every 24 hours.

SUMMARY:
Research studies raise the possibility that medications such as quetiapine may improve mood or reduce obsessions in people with anorexia nervosa and may even help to normalize appetite. The medication quetiapine also known as seroquel works by activating certain systems in the brain, such as ones known as dopamine and serotonin chemical systems in the brain.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18-65
* Must be at least 15% below ideal body weight

Exclusion Criteria:

* Allergy to quetiapine
* Diagnosis of schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-02; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine efficacy of seroquel in anorexia nervosa | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Floirda, Tampa, Florida, United States